CLINICAL TRIAL: NCT02229929
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Pharmacokinetics of Intravenous CR845 in Hemodialysis Patients, and Its Safety and Efficacy in Hemodialysis Patients With Uremic Pruritus
Brief Title: Safety and Pharmacokinetics of IV CR845 in Hemodialysis Patients, and Its Efficacy in Patients With Uremic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-CLIN2005
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Pruritus; Uremic Pruritus
Keywords: Pruritus; uremic pruritus; kappa opioid; CR845
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: Placebo (Placebo Comparator): Intravenous matched placebo
  Interventions: Drug: Part A: Placebo
- Part A: CR845 0.5 mcg/kg (Experimental): Intravenous CR845, 0.5 mcg/kg
  Interventions: Drug: Part A: CR845 0.5 mcg/kg
- Part A: CR845 1.0 mcg/kg (Experimental): Intravenous CR845, 1.0 mcg/kg
  Interventions: Drug: Part A: CR845 1.0 mcg/kg
- Part A: CR845 2.5 mcg/kg (Experimental): Intravenous CR845, 2.5 mcg/kg
  Interventions: Drug: Part A: CR845 2.5 mcg/kg
- Part B: Placebo (Placebo Comparator): Intravenous matched placebo
  Interventions: Drug: Part B: Placebo
- Part B: CR845 1.0 mcg/kg (Experimental): Intravenous CR845, 1.0 mcg/kg
  Interventions: Drug: Part B: CR845 1.0 mcg/kg

INTERVENTIONS:
Drug: Part A: Placebo — Part A: Single i.v. dose of Placebo administered after each dialysis session over a 1 week treatment period (3 times per week)
  Other Names: Matched Placebo
  Arms: Part A: Placebo
Drug: Part A: CR845 0.5 mcg/kg — Part A: Single i.v. dose of CR845 administered after each dialysis session over a 1 week treatment period (3 times per week)
  Other Names: CR845 0.5 mcg/kg
  Arms: Part A: CR845 0.5 mcg/kg
Drug: Part A: CR845 1.0 mcg/kg — Part A: Single i.v. dose of CR845 administered after each dialysis session over a 1 week treatment period (3 times per week)
  Other Names: CR845 1.0 mcg/kg
  Arms: Part A: CR845 1.0 mcg/kg
Drug: Part A: CR845 2.5 mcg/kg — Part A: Single i.v. dose of CR845 administered after each dialysis session over a 1 week treatment period (3 times per week)
  Other Names: CR845 2.5 mcg/kg
  Arms: Part A: CR845 2.5 mcg/kg
Drug: Part B: Placebo — Part B: Single i.v. dose of Placebo administered after each dialysis session over a 2 week treatment period (3 times per week)
  Other Names: Matched Placebo
  Arms: Part B: Placebo
Drug: Part B: CR845 1.0 mcg/kg — Part B: Single i.v. dose of CR845 administered after each dialysis session over a 2 week treatment period (3 times per week)
  Other Names: CR845 1.0 mcg/kg
  Arms: Part B: CR845 1.0 mcg/kg

SUMMARY:
The primary purpose of this study is to:

* Evaluate the safety and pharmacokinetic profile of repeated doses IV CR845 over one week in patients who are undergoing hemodialysis. (Part A)
* This study is also investigating whether repeated doses of IV CR845 over two weeks is safe and effective in reducing the intensity of itching in hemodialysis patients with uremic pruritus (Part B).

DETAILED DESCRIPTION:
Placebo-controlled

ELIGIBILITY:
Inclusion criteria:

* Able to provide written informed consent prior to any study procedures;
* Able to communicate clearly with the Investigator and staff, able to read and understand the study procedures;
* Males or females 18 years of age or older;
* End stage renal disease (ESRD) patients who have been on hemodialysis for at least three months and are currently on hemodialysis:

  * At least three times per week (Part A)
  * Three times per week (Part B)
* Has a body weight ≤ 135 kg
* Part B: Patient who self-reports daily or near daily pruritus during the 6 weeks prior to Screening;
* Part B: Patient who reports a Patient B or Patient C profile on the Patient Self-categorization of Pruritus Disease Severity questionnaire at Screening;
* Part B: At the end of the Run-in Period:

  * Patient who completed ratings of worst itching intensity [visual analog scale (VAS)] at least 8 times out of 14 VAS assessments;
  * Patient who has a mean value of >40 mm on the worst itching VAS over the one week Run-in Period.

Exclusion criteria:

* Known to be non-compliant with dialysis treatment (i.e., has a history of missed dialysis sessions due to non-compliance in the past 2 months);
* Anticipated to receive a kidney transplant during the study;
* Known history of allergic reaction to opiates such as hives (Note: side effects related to the use of opioids such as constipation or nausea would not exclude the patients from the study);
* Known or suspected history of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)-diagnosed alcohol, narcotic, or other drug abuse or dependence within 12 months prior to Screening;
* Acute or unstable medical condition(s) such as congestive heart failure [New York Heart Association (NYHA) class IV], which in the opinion of the Investigator would pose undue risk to the patient or would impede complete collection of the data or its evaluability;
* Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) greater than 2.5X the reference upper limit of normal (ULN), or bilirubin greater than 4X the ULN at Screening;
* Received another investigational drug within 30 days prior to the start of the Run-in Period or has planned to participate in another clinical trial while enrolled in this study
* Part B: Has pruritus probably or definitely attributed to a cause other than ESRD or its complications (e.g., patients with concomitant pruritic dermatological disease or cholestatic liver disease would be excluded). (Note: Patients whose pruritus is attributed to ESRD complications such as hyperparathyroidism, hyperphosphatemia, anemia, or the dialysis procedure or prescription may be enrolled);
* Part B: Has localized itch restricted to the palms of the hands as determined from the Brief Itch Inventory diagram, completed during the Screening Period;
* Part B: Has pruritus only during the dialysis session (by patient report);
* Part B: Has used gabapentin, calcineurin inhibitors, opioids; antipsychotics; systemic or topical corticosteroids (other than otic or ophthalmic preparations); sedatives; hypnotics; anti-anxiety agents selective serotonin reuptake inhibitors (SSRIs); or tricyclic antidepressants for < 4 weeks prior to the start of the Run-In Period or had a dose change within the previous 30 days;
* Part B: Is not willing to abstain from use of antihistamines (oral, IV, or topical) for 3 weeks (from the start of the Run-In Period through the end of Week 2);
* Part B: Not willing to abstain from making changes to topical non-drug treatments (e.g., emollients, creams, oils) for pruritus for 3 weeks (from the start of the Run-In Period through the end of Week 2);
* Part B: Received ultraviolet B treatment within 30 days prior to the start of the Run-in Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Part A: Determine the Pharmacokinetics of Repeated Doses of CR845 in Hemodialysis Patients (half-life, Cmax, Tmax, AUC, Vd) | 1 week
  To evaluate the pharmacokinetics of repeated doses of CR845 in hemodialysis patients over a one-week treatment period.
Part B: Change in Worst Itching Intensity using a 100-mm Visual Analog Scale | 2 weeks
  Change from baseline to the average of Week 2 worst itching (daytime and nighttime) VAS where 0 mm represents "No Itch" and 100 mm represents the "Worst Itch You Can Imagine".

SECONDARY OUTCOMES:
Part B: Change in quality-of-life assessed using the Skindex-10 survey | 2 weeks
  Change from baseline to Day 15 in itch-related quality of life as assessed by the total Skindex-10 scores
Part B: Sleep disturbance assessed using Itch Medical Outcomes Study (MOS) survey | 2 weeks
  Change from baseline to Day 15 in itch-related sleep disturbance based on the Itch MOS sleep problems index II (SLP-9)

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Menzaghi, PhD, Study Director — Cara Therapeutics, Inc.
Locations (20):
- United States (20):
  - US Renal Care, Pine Bluff, Arkansas
  - US Renal Care, Chula Vista, California
  - US Renal Care, Long Beach, California
  - Valley Renal Medical Group, Northridge, California
  - Nephrology Specialists Medical Group, Inc, Orange, California
  - North American Research Institute, San Dimas, California
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Emory Dialysis Center at Northside, Atlanta, Georgia
  - Western New England Renal & Transplant Associates, PC, Springfield, Massachusetts
  - US Renal Care, Gallup, New Mexico
  - Trude Weishaupt Memorial Dialysis Center, Fresh Meadows, New York
  - Winthrop University Hospital, Mineola, New York
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - US Renal Care, Aiken, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - US Renal Care, Grand Prairie, Texas
  - US Renal Care, San Antonio, Texas

REFERENCES:
- [Derived] Spencer RH, Noonan PK, Marbury T, Menzaghi F. Impact of renal impairment on the pharmacokinetic profile of intravenous difelikefalin, a kappa opioid receptor agonist for the treatment of pruritus. BMC Nephrol. 2024 Oct 14;25(1):351. doi: 10.1186/s12882-024-03790-w. PMID 39402448